CLINICAL TRIAL: NCT00448006
Title: A Clinical Feasibility Study to Evaluate the New Allium Biliary Stent, in Patients Suffering From "Malignant Biliary Duct Obstruction" (Endoscopic Insertion)
Brief Title: Clinical Feasibility Study of Allium's Biliary Stent
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Allium, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIS-CL-001
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2008-04

CONDITIONS: Malignant Obstruction of the Common Bile Duct
Keywords: common; bile; duct; biliary; malignant; obstruction; stent
MeSH Terms: conditions — Bites and Stings | interventions — Self Expandable Metallic Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Allium Biliary Stent — device
Device: allium biliary stent — allium biliary stent
  Other Names: self expandable stent

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Allium Biliary Stent in malignant obstructions of the common bile duct.

DETAILED DESCRIPTION:
Biliary duct stenoses are caused by intrinsic malignant disease of the common bile duct or by compression or infiltration of malignancies of the abdominal organs, i.e. pancreas, liver, stomach, duodenum, etc, or by iatrogenic reasons such as endoscopic biliary stone manipulations, biliary anastomoses or biliary duct reimplantation. In these diseases, a stent can be placed in the biliary duct canal to "open it" and relieve the obstruction. The Allium Biliary Stent is to be inserted into the biliary duct to allow free flow of biliary fluid from the liver to the duodenum by supporting the obstructed area of the biliary duct lumen, keep it open, and prevent its re-obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years or older
* Patient has malignant obstructive jaundice
* Patient is unfit for surgery
* Patient is capable of giving informed consent
* Patient is willing to comply with study requirements

Exclusion Criteria:

* Patient has a benign biliary duct obstruction
* Patient cannot tolerate any form of antibiotic treatment
* Patient is currently receiving anticoagulation therapy
* Patient has history of illness, medication, or surgery that may affect the efficacy of the stent (e.g.: a previous surgical change in the anatomy of the common bile duct)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04 (Estimated); Primary Completion 2009-08

PRIMARY OUTCOMES:
Body temperature measurement, patient comfort analysis, sonographic measurements of the duct channels, abdominal X-ray imaging of the stent, and blood tests will be performed at 24 hours, 30 days, 3, 6, and 12 months following stent insertion. | up to 12 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Simon Bar-Meir, M.D., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- See also: The Chaim Sheba Medical Center at Tel Hashomer — http://eng.sheba.co.il/main/siteNew/index.php